CLINICAL TRIAL: NCT04764669
Title: An Open-Label Study To Evaluate the Pharmacodynamic Effects, Efficacy, Safety, and Tolerability of E2027 in Subjects With Dementia With Lewy Bodies or Parkinson's Disease Dementia With or Without Amyloid Copathology
Brief Title: A Study of E2027 in Participants With Dementia With Lewy Bodies (DLB) or Parkinson's Disease Dementia (PDD) With or Without Amyloid Copathology
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2027-A001-203
Record Dates: First submitted 2021-02-19; First posted 2021-02-21 (Actual); Results first posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-08

CONDITIONS: Lewy Body Disease; Parkinson Disease
Keywords: E2027; Amyloid Copathology; Parkinson's Disease Dementia; Dementia With Lewy Bodies
MeSH Terms: conditions — Lewy Body Disease; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DLB Without Amyloid Copathology (Experimental): Participants with DLB (without amyloid copathology) will receive E2027 50 milligram (mg) capsules, orally, once daily up to 12 weeks.
  Interventions: Drug: E2027
- DLB With Amyloid Copathology (Experimental): Participants with DLB (with amyloid copathology) will receive E2027 50 mg capsules, orally, once daily up to 12 weeks.
  Interventions: Drug: E2027
- PDD Without Amyloid Copathology (Experimental): Participants with PDD (without amyloid copathology) will receive E2027 50 mg capsules, orally, once daily up to 12 weeks.
  Interventions: Drug: E2027
- PDD With Amyloid Copathology (Experimental): Participants with PDD (with amyloid copathology) will receive E2027 50 mg capsules, orally, once daily up to 12 weeks.
  Interventions: Drug: E2027

INTERVENTIONS:
Drug: E2027 — Oral hypromellose capsules.

SUMMARY:
The purpose of study is to demonstrate the pharmacodynamic (PD) effects of E2027 on cerebrospinal fluid (CSF) cyclic guanosine monophosphate (cGMP) in participants with DLB and PDD with and without amyloid copathology after 9 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 50 to 85 years, inclusive at time of consent
2. Meet criteria for probable DLB (as defined by the 4th report of the DLB Consortium) or meet criteria for probable PDD (as defined by the task force of the Movement Disorder Society).
3. Mini-mental state examination (MMSE) greater than (>) 14 and less than (<) 26 at Screening Visit
4. For DLB participants, have experienced visual hallucinations since onset of their DLB
5. If receiving acetylcholinesterase inhibitors (AChEIs), must have been on a stable dose for at least 12 weeks before Screening Visit, with no plans for dose adjustment during the study. Treatment naive participants can be entered into the study but there should be no plans to initiate treatment with AChEIs from Screening to the end of the study.
6. If receiving memantine, must have been on a stable dose for at least 12 weeks before Screening Visit, with no plans for dose adjustment during the study. Treatment naive participants can be entered into the study but there should be no plans to initiate treatment with memantine from Screening to the end of the study.
7. If receiving Parkinson's disease medications, must have been on a stable dose for at least 4 weeks before Screening Visit, with no plans for dose adjustment during the study.
8. Must have an identified caregiver or informant who is willing and able to provide follow up information on the participant throughout the course of the study.
9. Provide written informed consent.

Exclusion Criteria:

1. Any neurological condition that may be contributing to cognitive impairment above and beyond those caused by the participant's DLB or PDD, including any comorbidities detected by clinical assessment or magnetic resonance imaging (MRI) (identification of amyloid copathology is not exclusionary)
2. History of transient ischemic attacks or stroke within 12 months of Screening
3. Modified Hachinski Ischemic Scale >4
4. Parkinsonian (extrapyramidal) features with Hoehn and Yahr Scale (HYS) stage 4 or higher
5. Any major psychiatric diagnosis, including schizophrenia, bipolar disorder and current major depressive disorder as per Diagnostic and Statistical Manual of Mental Disorders Fifth Edition
6. Geriatric Depression Scale (GDS) score >8
7. Severe visual or hearing impairment that may interfere with the participant study assessments including cognitive testing
8. Any contraindications to lumbar puncture
9. History of deep brain stimulation or other neurosurgical procedure for Parkinson's disease
10. Has thyroid stimulating hormone (TSH) above normal range
11. Abnormally low serum vitamin B12 levels (< the lower limit of normal [LLN]) for the testing laboratory
12. Contraindications to MRI scanning
13. Evidence of other clinically significant lesions that suggest a dementia diagnosis other than DLB or PDD on brain MRI at Screening
14. Other significant pathological findings on brain MRI at Screening
15. Hypersensitivity to E2027 or any of the excipients
16. A prolonged corrected QT interval calculated using Fridericia's formula (QTcF) as demonstrated by triplicate ECG at the Screening or Baseline Visit (that is, mean value >450 millisecond [msec])
17. Had symptomatic orthostatic hypotension or symptomatic orthostatic tachycardia which resulted in hospitalization or urgent medical review in hospital in the past 12 months before Screening
18. Any other clinically significant abnormalities in vital signs, ECG and laboratory values that in the opinion of the investigator, require further investigation or treatment or that may interfere with study procedures or safety
19. Malignant neoplasms within 3 years of Screening (except for basal or squamous cell carcinoma of the skin, or localized prostate cancer in male participants). Participants who had malignant neoplasms but who have had at least 3 years of documented uninterrupted remission before Screening need not be excluded.
20. Has a "yes" answer to C-SSRS suicidal ideation Type 4 or 5, or any suicidal behavior assessment within 6 months before Screening, at Screening, or at the Baseline Visit, or has been hospitalized or treated for suicidal behavior in the past 5 years before Screening
21. Known or suspected history of drug or alcohol dependency or abuse within 2 years before Screening, current use of recreational drugs or a positive urine drug test at Screening.
22. Any other medical conditions (example, cardiac, respiratory, gastrointestinal, renal disease) which are not stably and adequately controlled, or which in the opinion of the investigator may affect the participant's safety or interfere with the study assessments
23. Taking any of the prohibited medications or not meeting the requirements regarding stable doses of permitted medications
24. Participation in a clinical study involving any investigational drug/device for DLB or PDD within 6 months before Screening or any other investigational drug/device in the 8 weeks or 5 half-lives (whichever is longer) of the study medication before Screening unless it can be documented that the participant was in a placebo treatment arm
25. Planned surgery which requires general, spinal or epidural anesthesia that will take place during the study.
26. Males who have not had a successful vasectomy (confirmed azoospermia) if their female partners are of childbearing potential and are not willing to use a highly effective contraceptive method throughout the study period and for 98 days after study drug discontinuation. No sperm donation is allowed during the study period and for 98 days after study drug discontinuation.
27. Females who are breastfeeding or pregnant at Screening or Baseline
28. Females of childbearing potential who:

    * Within 28 days before study entry, did not use a highly effective method of contraception
    * Do not agree to use a highly effective method of contraception throughout the entire study period and for 28 days after study drug discontinuation

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2021-12-08 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (13):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - JEM Research Institute, Atlantis, Florida
  - Elias Research Associates (Allied Biomedical Research Institute), Miami, Florida
  - Napa Research, Pompano Beach, Florida
  - University of South Florida, Department of Psychiatry and Behavioral Neurosciences, Tampa, Florida
  - Alzheimer's Research and Treatment Center, Wellington, Florida
  - University of Kentucky, Dept of Neurology, Sanders Brown Center on Aging, Lexington, Kentucky
  - Advanced Memory Research Institute of NJPC, Toms River, New Jersey
  - Neurological Associates of Albany, PC, Albany, New York
  - Columbia University Medical Center, New York, New York
  - Neurology Diagnostics, Inc., Dayton, Ohio
  - Cleveland Clinic, Lou Ruvo Center for Brain Health at Lakewood Hospital, Lakewood, Ohio
  - Summit Research Network (Oregon) Inc., Portland, Oregon
- Toronto Memory Program, Toronto, Canada

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 15 investigative sites in the United States, and Canada from 25 Feb 2021 to 27 Jan 2022.
Pre-assignment Details: A total of 83 participants were screened, of which 49 were screen failures and 34 participants received the study treatment.
Groups:
- DLB Without Amyloid Copathology: Participants with dementia with Lewy bodies (DLB) (without amyloid copathology) received E2027 50 milligram (mg) capsules, orally, once daily up to 12 weeks.
- DLB With Amyloid Copathology: Participants with DLB (with amyloid copathology) received E2027 50 mg capsules, orally, once daily up to 12 weeks.
- PDD Without Amyloid Copathology: Participants with Parkinson's Disease Dementia (PDD) (without amyloid copathology) received E2027 50 mg capsules, orally, once daily up to 12 weeks.
- PDD With Amyloid Copathology: Participants with PDD (with amyloid copathology) received E2027 50 mg capsules, orally, once daily up to 12 weeks.
Period: Overall Study
Arm/Group | DLB Without Amyloid Copathology | DLB With Amyloid Copathology | PDD Without Amyloid Copathology | PDD With Amyloid Copathology
Started | 10 | 11 | 10 | 3
Completed | 7 | 11 | 8 | 3
Not Completed | 3 | 0 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Subject Choice | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included participants who received at least 1 dose of study drug and had at least 1 post baseline safety assessment.
Groups:
- DLB Without Amyloid Copathology: Participants with DLB (without amyloid copathology) received E2027 50 mg capsules, orally, once daily up to 12 weeks.
- PDD Without Amyloid Copathology: Participants with PDD (without amyloid copathology) received E2027 50 mg capsules, orally, once daily up to 12 weeks.
- Total: Total of all reporting groups
Arm/Group | DLB Without Amyloid Copathology | DLB With Amyloid Copathology | PDD Without Amyloid Copathology | PDD With Amyloid Copathology | Total
Number analyzed (Participants) | 10 | 11 | 10 | 3 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.2 (6.21) | 73.9 (6.07) | 74.4 (6.40) | 78.3 (2.52) | 73.9 (6.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 1 | 13
  Male | 6 | 8 | 5 | 2 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 1 | 3
  Not Hispanic or Latino | 9 | 11 | 9 | 2 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 10 | 11 | 9 | 3 | 33
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Cerebrospinal Fluid (CSF) Cyclic Guanosine Monophosphate (cGMP) at Week 9
Description: cGMP was measured in CSF samples using a validated liquid chromatography with tandem mass spectrometry (LC-MS/MS) method with a lower limit of quantitative at 0.500 nanogram per milliliter (ng/ml). Evaluation of cGMP following dosing of E2027 was based on relative percent change from baseline.
Time Frame: Baseline, Week 9
Population: Pharmacodynamic (PD) analysis set included participants who had sufficient PD data to derive at least 1 PD parameter.
Measure: Least Squares Mean (Standard Error); unit: Percent Change in CSF (ng/mL)
Arm/Group | DLB Without Amyloid Copathology | DLB With Amyloid Copathology | PDD Without Amyloid Copathology | PDD With Amyloid Copathology
Number analyzed (Participants) | 9 | 10 | 10 | 3
Percent Change in CSF (ng/mL) | 230.412 (20.417) | 250.434 (17.015) | 186.869 (24.374) | 362.519 (40.764)
Statistical Analysis 1: Comparison: DLB Without Amyloid Copathology vs DLB With Amyloid Copathology; Test type: Superiority — Primary comparisons were: DLB without amyloid copathology versus DLB with amyloid copathology; Least squares mean difference = -20.022, 95% CI 2-sided [-77.635 to 37.591]
Statistical Analysis 2: Comparison: PDD Without Amyloid Copathology vs PDD With Amyloid Copathology; Test type: Superiority — Primary comparisons were: PDD without amyloid copathology versus PDD with amyloid copathology; Least squares mean difference = -175.650, 95% CI 2-sided [-287.407 to -63.893]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Severe TEAEs, Serious TEAEs, Adverse Events (AEs) Resulting in Study Discontinuation
Description: A TEAE was defined as an AE that emerged during treatment, having been absent at pretreatment or reemerged during treatment, having been present at pretreatment but stopped before treatment, or worsened in severity during treatment relative to the pretreatment state, when the AE is continuous. Severe TEAE was defined as inability to work or to perform normal daily activity. A Serious TEAE was any untoward medical occurrence that at any dose: resulted in death; life threatening condition; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect or was medically important due to other reasons than the above mentioned criteria. An AE was defined as any untoward medical occurrence in a participant administered an investigational product. AE resulting in study discontinuation was defined as AE due to which the study medication was stopped.
Time Frame: From first dose of study drug up to Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | DLB Without Amyloid Copathology | DLB With Amyloid Copathology | PDD Without Amyloid Copathology | PDD With Amyloid Copathology
Number analyzed (Participants) | 10 | 11 | 10 | 3
Participants
  TEAEs | 6 | 4 | 3 | 2
  Severe TEAEs | 1 | 0 | 0 | 0
  Serious TEAEs | 1 | 0 | 0 | 0
  AE Leading to Discontinuation from Study | 1 | 0 | 1 | 0

3. Secondary Outcome: Number of Participants With Treatment Emergent Orthostatic Hypotension
Description: Orthostatic hypotension was defined based on the following criteria per protocol: Drop in standing systolic blood pressure (SBP) greater than or equal to (>=) 20 millimeter of mercury (mmHg) compared to supine or drop in standing diastolic blood pressure (DBP) >=10 mmHg compared to supine. Treatment-emergent orthostatic hypotension was defined as: if at baseline participant did not have SBP drop >=20 mmHg and no DBP drop >=10 mmHg, but developed one or more of these two events during post baseline visits.
Time Frame: Week 3, Week 6, Week 9, Week 12 and Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | DLB Without Amyloid Copathology | DLB With Amyloid Copathology | PDD Without Amyloid Copathology | PDD With Amyloid Copathology
Number analyzed (Participants) | 10 | 11 | 10 | 3
Participants
  Week 3 | 0 | 1 | 1 | 0
  Week 6 | 0 | 3 | 1 | 0
  Week 9 | 2 | 1 | 1 | 0
  Week 12 | 0 | 3 | 2 | 0
  Week 16 | 1 | 3 | 1 | 0

4. Secondary Outcome: Number of Participants With Post Baseline Treatment Emergent Orthostatic Tachycardia
Description: Orthostatic tachycardia was defined by the following criteria per protocol: Standing heart rate (HR) increased by greater than (>) 30 beats/min compared to supine and absolute standing HR was >100 beats/min. A participant was counted as treatment-emergent if orthostatic tachycardia emerged during the treatment, having been absent at baseline (pretreatment).
Time Frame: From first dose of study drug up to Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | DLB Without Amyloid Copathology | DLB With Amyloid Copathology | PDD Without Amyloid Copathology | PDD With Amyloid Copathology
Number analyzed (Participants) | 10 | 11 | 10 | 3
Participants | 0 | 1 | 0 | 0

5. Secondary Outcome: Number of Participants With Markedly Abnormal Laboratory Values
Description: A laboratory value was determined to be a markedly abnormal value if the postbaseline grade increased from baseline and the post-baseline grade was greater than or equal to 2. Markedly abnormal laboratory values were based on Common Terminology Criteria for Adverse events (CTCAE) Version 5.0.
Time Frame: From first dose of study drug up to Week 16
Population: Safety analysis set included participants who received at least 1 dose of study drug and had at least 1 post baseline safety assessment. Number analyzed "n" are the participants who were evaluable for the outcome measure for given categories.
Measure: Count of Participants; unit: Participants
Arm/Group | DLB Without Amyloid Copathology | DLB With Amyloid Copathology | PDD Without Amyloid Copathology | PDD With Amyloid Copathology
Number analyzed (Participants) | 10 | 11 | 10 | 3
Participants
  Creatinine: Markedly Abnormal High: number analyzed (Participants) | 10 | 11 | 9 | 3
  Creatinine: Markedly Abnormal High | 0 | 0 | 0 | 2
  Lymphocytes: Markedly Abnormal Low: number analyzed (Participants) | 10 | 11 | 9 | 3
  Lymphocytes: Markedly Abnormal Low | 0 | 0 | 0 | 1
  Potassium: Markedly Abnormal High: number analyzed (Participants) | 10 | 11 | 9 | 3
  Potassium: Markedly Abnormal High | 0 | 0 | 1 | 0

6. Secondary Outcome: Number of Participants With Post-Baseline Abnormal Electrocardiogram (ECG) Findings
Description: Abnormal ECG findings were defined as follows: corrected QT interval calculated using Fridericia's formula (QTcF) prolonged by >60 millisecond (ms) from baseline and absolute QTcF >450 ms; QTcF prolonged to >500 ms; Change from baseline of PR interval >=25 percent (%) to an absolute PR value of >220 ms; Change from baseline of QRS interval >=25% to an absolute QRS value of >120 ms.
Time Frame: From first dose of study drug up to Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | DLB Without Amyloid Copathology | DLB With Amyloid Copathology | PDD Without Amyloid Copathology | PDD With Amyloid Copathology
Number analyzed (Participants) | 10 | 11 | 10 | 3
Participants
  QTcF prolongation by >60 ms from baseline and absolute QTcF >450 ms | 0 | 0 | 0 | 0
  QTcF prolonged to >500 ms | 0 | 0 | 0 | 0
  Change from baseline of PR >= 25% to an absolute PR value of >220 msec | 0 | 0 | 0 | 0
  Change from baseline of QRS >= 25% to an absolute QRS value of >120 msec | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Suicidal Ideation or Suicidal Behavior as Measured Using Columbia Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS (mapped to Columbia Classification Algorithm of Suicide Assessment (C-CASA) categories); is an interview-based instrument to systematically assess suicidal ideation and suicidal behavior. C-SSRS assess whether participant experience any of the following: completed suicide; suicide attempt (response of "yes" on "actual attempt"); preparatory acts toward imminent suicidal behavior ("yes" on "preparatory acts or behavior", "aborted attempt" or "interrupted attempt"), suicidal ideation ("yes" on "wish to be dead", "non-specific active suicidal thoughts", "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent, any self-injurious behavior with no suicidal intent ("yes" on "has participant engaged in non-suicidal self-injurious behavior"). Here, number of participants with positive response ("yes") to suicidal behavior or/and Ideation, any non-suicidal self-injurious behavior was reported.
Time Frame: From first dose of study drug up to Week 16
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | DLB Without Amyloid Copathology | DLB With Amyloid Copathology | PDD Without Amyloid Copathology | PDD With Amyloid Copathology
Number analyzed (Participants) | 10 | 11 | 10 | 3
Participants
  Completed Suicide | 0 | 0 | 0 | 0
  Suicide Attempt | 0 | 0 | 0 | 0
  Preparatory Actions Towards Imminent Suicidal Behavior | 0 | 0 | 0 | 0
  Wish to Die | 0 | 0 | 0 | 0
  Actual Suicidal Thoughts; Non-specific | 0 | 0 | 0 | 0
  Actual Suicidal Thoughts with Method; No Intent | 0 | 0 | 0 | 0
  Active Thoughts with Intent | 0 | 0 | 0 | 0
  Active Thoughts with Plan and Intent | 0 | 0 | 0 | 0
  Self-injurious Behavior; No Intent | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Total Score of Unified Parkinson's Disease Rating Scale Part III: Motor Examination (UPDRS-III)
Description: The UPDRS scale evaluates extrapyramidal features in motor function in Parkinson's disease. It contains 33 items in 18 categories: (1) speech, (2) facial expression, (3) rigidity, (4) finger tapping, (5) hand movements, (6) supinational and pronation movements of hands, (7) toe tapping, (8) leg agility, (9) arising from chair, (10) gait, (11) freezing of gait, (12) postural stability, (13) posture, (14) body bradykinesia, (15) postural tremor of hands, (16) kinetic tremor of hands, (17) rest tremor amplitude and (18) constancy of rest tremor. Each item is scored 0 to 4, giving a total score range 0 to 132. Higher scores indicating more severe symptoms.
Time Frame: Baseline, Week 12 and Week 16
Population: Safety analysis set included participants who received at least 1 dose of study drug and had at least 1 post baseline safety assessment. Here number analyzed "n" are the participants who were evaluable for the outcome measure for given time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DLB Without Amyloid Copathology | DLB With Amyloid Copathology | PDD Without Amyloid Copathology | PDD With Amyloid Copathology
Number analyzed (Participants) | 10 | 11 | 10 | 3
score on a scale
  Baseline | 21.1 (9.81) | 24.6 (12.33) | 28.9 (12.35) | 38.0 (19.00)
  Change at Week 12: number analyzed (Participants) | 9 | 11 | 9 | 3
  Change at Week 12 | 5.0 (4.61) | 6.5 (7.20) | 2.8 (10.67) | -4.0 (5.29)
  Change at Week 16: number analyzed (Participants) | 7 | 11 | 9 | 3
  Change at Week 16 | 1.1 (13.92) | 2.1 (8.01) | 4.3 (17.01) | 2.3 (2.31)

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 16
Arm/Group | DLB Without Amyloid Copathology | DLB With Amyloid Copathology | PDD Without Amyloid Copathology | PDD With Amyloid Copathology
All-Cause Mortality (participants affected / at risk) | 1/10 | 0/11 | 0/10 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/11 | 0/10 | 0/3
Other Adverse Events (participants affected / at risk) | 5/10 | 4/11 | 3/10 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DLB Without Amyloid Copathology (N=10) | DLB With Amyloid Copathology (N=11) | PDD Without Amyloid Copathology (N=10) | PDD With Amyloid Copathology (N=3)
Death (General disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DLB Without Amyloid Copathology (N=10) | DLB With Amyloid Copathology (N=11) | PDD Without Amyloid Copathology (N=10) | PDD With Amyloid Copathology (N=3)
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Temperature intolerance (General disorders) | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Aggression (Psychiatric disorders) | 1 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Due to insufficient numbers enrolled of participants with PDD and amyloid copathology, interpretation of results in this subgroup is limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT04764669/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT04764669/SAP_001.pdf